CLINICAL TRIAL: NCT06303037
Title: Determination of the 95% Effective Dose of Remimazolam in Combination With Different Doses of Esketamine During Gastroscopy in Children
Brief Title: Effect of Esketamine on 95% Induction Dose of Remimazolam
Acronym: EEIDR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2024-03-105
Record Dates: First submitted 2024-01-25; First posted 2024-03-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pediatric; Gastroscopy; ED95; Sedation
Keywords: remimazolam; esketamine
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Experimental): Low-dose esketamine
  Interventions: Drug: Remimazolam besylate and low-dose Esketamine
- Group M (Experimental): Medium dose esketamine
  Interventions: Drug: Remimazolam besylate and Medium dose Esketamine

INTERVENTIONS:
Drug: Remimazolam besylate and low-dose Esketamine — Esketamine was injected intravenously 0.25mg/kg and the initial dose of Remimazolam was 0.3mg/kg
  Other Names: intravenous bolus remimazolam according to biased coin design
  Arms: Group L
Drug: Remimazolam besylate and Medium dose Esketamine — Esketamine was injected intravenously 0.5mg/kg and the initial dose of Remimazolam was 0.2mg/kg
  Other Names: intravenous bolus remimazolam according to biased coin design
  Arms: Group M

SUMMARY:
As an invasive operation, gastroscopy will cause children's nervousness, anxiety and uncooperative behavior, and even lead to the risk of bleeding and perforation, which will also affect the accuracy of the examination results.The purpose of this study is to explore the influence of different doses of esketamine on the induced dose ED95 of remazolam during gastroscopic placement in children, and to provide theoretical basis for the combined use of remimazolam besylate and esketamine in gastroscopic anesthesia in children.

DETAILED DESCRIPTION:
Children aged 3-12 who underwent gastroscopy were randomly divided into two groups: L group with Esketamine 0.25mg/kg and the initial dose of Remimazolam was 0.3mg/kg ,M group with Esketamine 0.5mg/kg and the initial dose of Remimazolam was 0.2mg/kg.Judging whether the sedation level of the children can meet the requirements of gastroscopy placement after injecting Remimazolam.The next dose was adjusted to 0.05mg/kg according to biased coin design,to further explore the induced dose of ED95 of Remimazolam under the background of different doses of Esketamine.

ELIGIBILITY:
Inclusion Criteria:

1. with American Society of Anesthesiologists (ASA) physical status I or II#;
2. aged 3#12 years#;
3. children with weight for age within the normal range#;
4. were scheduled to have a gastroscopy;

Exclusion Criteria:

1. Children who had gastrointestinal,Cardiovascular or endocrine dysfunction;
2. contraindication to preoperative sedation or had a known allergy or hypersensitive reaction to remimazolam and esketamine;
3. recently respiratory infection, mental disorder;
4. other reasons that researchers hold it is not appropriate to participate in this trial.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Sedation induction time | during anaesthetic induction
  the patients' unresponsiveness to the mild shaking of their shoulder

SECONDARY OUTCOMES:
Modified observer's assessment of alertness#sedation#MOAA/S#scale | 1 minutes after single intravenous bolus remimazolam
  5#Subject responds readily to name spoken in a normal tone; 4 #Lethargic response of a subject to a name spoken in a normal tone; 3 #The subject responds only after a name is called loudly and repeatedly; 2 #The subject responds only after mild prodding or shaking;
  1 #The subject responds only after a painful trapezius squeeze; 0 #The subject does not respond to painful trapezius squeeze. MOAA/S score ≤ 2 points represent successful sedation
Recovery times | Within up to 30 minutes after operation
  The time from discontinuation of anesthesia drug to the first open eye of the children and to achieve aldrete≥9
VAS(The difficulty of gastroscope insertion) | Moment of endoscopic insertion
  VAS values range from 0 to 10. A value of 0 represents that gastroscopy placement is very easy.and 10 represents that gastroscopy placement is very difficult.
Number of children with adverse effects | Within 24 hours after completion of gastroscopy.
  Bradycardia and/or hypotension need for hemodynamic support Desaturation is defined as Oxygen desaturation <90% Any adverse effects requiring interventions

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Yuhang Cai, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Qiaoqiao Wang, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China